CLINICAL TRIAL: NCT00984360
Title: A Pilot Trial of Naltrexone for Methamphetamine Addiction - Role of the A118G SNP
Brief Title: Study of Naltrexone for Methamphetamine Addiction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, John Mendelson, MD, Senior Scientist, California Pacific Medical Center Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DA027161-01 (NIH)
Record Dates: First submitted 2009-09-14; First posted 2009-09-25 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Methamphetamine Dependence
Keywords: Meth; Methamphetamine Addiction; Methamphetamine Treatment; Naltrexone; Vivitrol; A118G; OPRM1
MeSH Terms: interventions — Naltrexone; vivitrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A118G (Experimental)
  Interventions: Drug: Naltrexone
- Wild-type (Experimental)
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — 380mg extended-release, given once by intramuscular gluteal injection
  Other Names: Vivitrol; Vivitrex

SUMMARY:
The purpose of this study is to determine whether methamphetamine-dependent individuals will use less methamphetamine when treated with naltrexone. The study will also investigate whether individuals with the mu opioid receptor gene variant A118G will use less methamphetamine than individuals without A118G.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* Patient is agreeable to conditions of study and signs consent form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
MA (-) Urine Samples | Twice weekly for 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Mendelson, MD, Principal Investigator — California Pacific Medical Center
Locations (1):
- Addiction & Pharmacology Research Laboratory, San Francisco, California, United States